CLINICAL TRIAL: NCT01323673
Title: Ethanol-Free Clobetasol Propionate Foam 0.05% (Olux-E Foam) vs Vehicle Foam in the Treatment of Chronic Hand Dermatitis.
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Stiefel, a GSK Company (Industry)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Organization: GlaxoSmithKline (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 115054
Record Dates: First submitted 2011-03-24; First posted 2011-03-25 (Estimated); Results first posted 2011-12-21 (Estimated); Last update posted 2018-06-20 (Actual); Status verified 2018-06

CONDITIONS: Dermatitis, Chronic
MeSH Terms: conditions — Dermatitis; Bronchiolitis Obliterans Syndrome

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Clobetasol Propionate 0.05% (Active Comparator)
  Interventions: Drug: clobetasol propionate 0.05%
- Vehicle (Placebo Comparator)
  Interventions: Drug: Vehicle / Placebo

INTERVENTIONS:
Drug: clobetasol propionate 0.05% — 2 times a day, 14 total days study treatment
  Arms: Clobetasol Propionate 0.05%
Drug: Vehicle / Placebo — 2 times a day, 14 total days of study treatment
  Arms: Vehicle

SUMMARY:
The purpose of this study is to determine how clobetasol proprionate foam works against a placebo foam in the treatment of hand dermatitis.

DETAILED DESCRIPTION:
Topical corticosteroids have anti-inflammatory, immunosuppressive and antiproliferative properties. Clobetasol propionate foam 0.05% (Olux-E), a Class 1 corticosteroid, is formulated in an ethanol free petrolatum base that provides the benefits of a super-potent corticosteroid combined with moisturizing ingredients in the treatment of corticosteroid responsive dermatoses. The current study is designed to show efficacy and safety in the treatment of moderate to severe chronic hand dermatitis.

ELIGIBILITY:
Inclusion Criteria:

* Capable of understanding and willing to provide signed informed consent
* Male or female at least 12 years of age at time of consent and at time of first dose.
* Able to complete the study and to comply with study instructions.
* Moderate to severe hand dermatitis.
* Chronic hand dermatitis diagnosis must be at least 6 months

Exclusion Criteria:

* Female who is pregnant, trying to become pregnant, or breast feeding.
* Currently diagnosed with allergic contact dermatitis.
* Participated in a previous study of the same study product.
* Had any major illness within 30 days before the screening/baseline visit.
* Considered immunocompromised.
* Has a clinically relevant history of or current evidence of abuse of alcohol or other drugs.
* Considered unable or unlikely to attend the necessary visits.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 125 (Actual)
Dates: Start 2010-11-15; Primary Completion 2011-03-01 (Actual); Study Completion 2011-03-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (9):
- United States (9):
  - GSK Investigational Site, San Diego, California
  - GSK Investigational Site, Boynton Beach, Florida
  - GSK Investigational Site, West Palm Beach, Florida
  - GSK Investigational Site, Louisville, Kentucky
  - GSK Investigational Site, Belleville, New Jersey
  - GSK Investigational Site, Montclair, New Jersey
  - GSK Investigational Site, Knoxville, Tennessee
  - GSK Investigational Site, Nashville, Tennessee
  - GSK Investigational Site, Austin, Texas

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Derived] Kircik LH, Eastman WJ, Gwazdauskas J. A randomized, double-blind phase 4 study of the efficacy and safety of ethanol-free clobetasol propionate foam, 0.05%, vs vehicle foam in the treatment of chronic hand dermatitis. J Drugs Dermatol. 2013 Mar;12(3):328-34. PMID 23545917
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Dataset Specification: 115054 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 115054 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 115054 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 115054 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 115054 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 115054 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 115054 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Groups:
- Olux-E Foam: Olux-E foam containing 0.05% clobestasol propionate, applied twice daily (morning and evening [BD]) for two weeks using the smallest amount of study product necessary to cover all affected areas, up to a maximum dosage of 50 grams (g) per week
- Vehicle Foam: Vehicle foam without the active ingredient clobestasol propionate, applied BD for two weeks using the smallest amount of study product necessary to cover all affected areas, up to a maximum dosage of 50 g per week
Period: Overall Study
Arm/Group | Olux-E Foam | Vehicle Foam
Started | 62 | 63
Completed | 59 | 58
Not Completed | 3 | 5
Not completed — Adverse Event | 0 | 1
Not completed — Lost to Follow-up | 0 | 1
Not completed — Protocol Violation | 1 | 0
Not completed — Withdrawal by Subject | 2 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Olux-E Foam | Vehicle Foam | Total
Number analyzed (Participants) | 62 | 63 | 125
Age, Continuous [Mean (Standard Deviation); unit: Years] | 51.5 (16.4) | 47.3 (14.3) | 49.4 (15.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 41 | 29 | 70
  Male | 21 | 34 | 55
Race/Ethnicity, Customized [Number; unit: participants]
  American Indian or Alaska Native | 2 | 2 | 4
  Asian | 1 | 2 | 3
  Black | 9 | 7 | 16
  Multiracial | 1 | 2 | 3
  White | 49 | 50 | 99

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Improvement of at Least 2 Grades in the Investigator's Static Global Assessment (ISGA) (Target Hand) Score From Baseline to Day 15
Description: The investigator rated chronic hand dermatitis of the participants' target hand using the 5-point ISGA: 0=clear, minor residual discoloration, no erythema (redness of skin)/induration (skin hardening)/papulation (eruption of small, rounded solid bumps on skin), no oozing/crusting; 1=almost clear, trace faint pink erythema, no induration/papulation and no oozing/crusting; 2=mild, faint pink erythema, mild induration/papulation; 3=moderate, pink-red erythema, moderate induration/papulation, some oozing/crusting; 4=Severe, bright-red erythema, severe induration/papulation, oozing/crusting.
Time Frame: Baseline (Day 1) and Day 15
Population: Intent-to-Treat (ITT) Population: all randomized participants who were dispensed study product. Missing values were imputed using last observation carried forward (LOCF, i.e., the last available observation, including Baseline, for a participant was used to estimate subsequent missing data points).
Measure: Number; unit: participants
Arm/Group | Olux-E Foam | Vehicle Foam
Number analyzed (Participants) | 62 | 63
participants | 26 | 18
Statistical Analysis 1: Comparison: Olux-E Foam vs Vehicle Foam; Test type: Superiority or Other; p = 0.151, Cochran-Mantel-Haenszel — Cochran-Mantel-Haenszel (CMH) test stratified by center was used for analysis

2. Secondary Outcome: Number of Participants With an Improvement of at Least 1 Grade in the ISGA (Target Hand) Score From Baseline to Day 15
Description: as for outcome 1
Time Frame: Baseline (Day 1) and Day 15
Population: ITT Population. Missing values were imputed using LOCF (i.e., the last available observation, including Baseline, for a participant was used to estimate subsequent missing data points).
Measure: Number; unit: participants
Arm/Group | Olux-E Foam | Vehicle Foam
Number analyzed (Participants) | 62 | 63
participants | 45 | 38

3. Secondary Outcome: Number of Participants With an Improvement of at Least 2 Grades in the ISGA (Target Hand) Score From Baseline to Day 3 and to Day 8
Description: as for outcome 1
Time Frame: Baseline (Day 1), Day 3, and Day 8
Population: as for outcome 2
Measure: Number; unit: participants
Arm/Group | Olux-E Foam | Vehicle Foam
Number analyzed (Participants) | 62 | 63
participants
  Day 3 | 2 | 3
  Day 15 | 12 | 11

4. Secondary Outcome: Number of Participants With an Improvement of at Least 1 Grade in the ISGA (Target Hand) Score From Baseline to Day 3 and and to Day 8
Description: as for outcome 1
Time Frame: Baseline (Day 1), Day 3, and Day 8
Population: as for outcome 2
Measure: Number; unit: participants
Arm/Group | Olux-E Foam | Vehicle Foam
Number analyzed (Participants) | 62 | 63
participants
  Day 3 | 24 | 14
  Day 8 | 36 | 32

5. Secondary Outcome: Number of Participants With an ISGA (Target Hand) Score of 0 or 1 at Days 3, 8, and 15
Description: as for outcome 1
Time Frame: Days 3, 8, and 15
Population: as for outcome 2
Measure: Number; unit: participants
Arm/Group | Olux-E Foam | Vehicle Foam
Number analyzed (Participants) | 62 | 63
participants
  Day 3 | 2 | 2
  Day 8 | 11 | 9
  Day 15 | 24 | 17

6. Secondary Outcome: Number of Participants With an Improvement of at Least 1 Grade in the Subject Global Assessment (SGA) (Target Hand) Score From Baseline to Days 3, 8, and 15
Description: On Days 1, 3, 8, and 15 prior to the investigator assessment, participants rated chronic hand dermatitis of the target hand using the 5-point SGA: 0=skin is clear; 1=dermatitis in minimal, there may be a few light-pink areas; 2=dermatitis is mild, there may be occasional light-pink areas; 3=dermatitis is moderate, there may be easily noticeable pink-red areas; 4=dermatitis is severe, there may be deep or bright-red areas that may be warm to the touch.
Time Frame: Baseline (Day 1) and Days 3, 8, and 15
Population: as for outcome 2
Measure: Number; unit: participants
Arm/Group | Olux-E Foam | Vehicle Foam
Number analyzed (Participants) | 62 | 63
participants
  Day 3 | 28 | 25
  Day 8 | 44 | 35
  Day 15 | 51 | 33

7. Secondary Outcome: Number of Participants With an SGA (Target Hand) Score of 0 or 1 at Days 3, 8, and 15
Description: as for outcome 6
Time Frame: Days 3, 8, and 15
Population: as for outcome 2
Measure: Number; unit: participants
Arm/Group | Olux-E Foam | Vehicle Foam
Number analyzed (Participants) | 62 | 63
participants
  Day 3 | 7 | 4
  Day 8 | 16 | 10
  Day 15 | 32 | 14

8. Secondary Outcome: Percent Change From Baseline in Pruritus, Stinging, Burning, and Pain Scores (Target Hand) at Days 3, 8, and 15
Description: On Days 1, 3, 8, and 15, participants assessed the pruritis (itching), stinging (piercing pain), burning, and pain of the target hand. Participants were instructed to assess the level/severity of the indicated symptoms over the previous 24 hours using a scale ranging from 0 (none) to 10 (unbearable). Percent change from baseline was calculated as value at Days 3, 8, and 15 minus the value at Baseline divided by the Baseline value * 100.
Time Frame: Baseline (Day 1) and Days 3, 8, and 15
Population: ITT Population. Only those participants contributing data at the indicated time points were analyzed.
Measure: Mean (Standard Deviation); unit: Percent change in scores on a scale
Arm/Group | Olux-E Foam | Vehicle Foam
Number analyzed (Participants) | 60 | 60
Percent change in scores on a scale
  Pruritus, Day 3, n=58, 58 | -29.4 (38.66) | -11.5 (52.76)
  Pruritus, Day 8, n=57, 57 | -48.3 (46.38) | -20.3 (62.98)
  Pruritus, Day 15, n=60, 59 | -65.7 (38.25) | -25.3 (58.18)
  Stinging, Day 3, n=57, 60 | -27.8 (37.86) | -1.84 (85.43)
  Stinging, Day 8, n=56, 58 | -49.2 (47.25) | -22.9 (59.17)
  Stinging, Day 15, n=58, 59 | -63.1 (40.63) | -28.9 (48.48)
  Burning, Day 3, n=57, 59 | -26.4 (40.77) | -10.4 (84.39)
  Burning, Day 8, n=55, 58 | -49.7 (49.87) | -26.1 (61.75)
  Burning, Day 15, n=59, 60 | -63.2 (45.46) | -31.1 (55.67)
  Pain, Day 3, n=56, 58 | -22.9 (54.80) | -21.0 (81.02)
  Pain, Day 8, n=57, 56 | -40.2 (52.25) | -21.5 (76.75)
  Pain, Day 15, n=60, 59 | -60.6 (41.76) | -35.5 (57.54)

ADVERSE EVENTS:
Arm/Group | Olux-E Foam | Vehicle Foam
Serious Adverse Events (participants affected / at risk) | 0/62 | 0/63
Other Adverse Events (participants affected / at risk) | 11/62 | 5/63
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Olux-E Foam (N=62) | Vehicle Foam (N=63)
Conjunctivitis (Eye disorders) | 0 | 1
Abdominal Pain Upper (Gastrointestinal disorders) | 1 | 0
Diarrhea (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0
Application Site Pruritus (General disorders) | 1 | 0
Nasopharyngitis (Infections and infestations) | 3 | 1
Sinusitis (Infections and infestations) | 1 | 1
Upper Respiratory Tract Infection (Infections and infestations) | 1 | 0
Skin Laceration (Injury, poisoning and procedural complications) | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Musculoskeletal Stiffness (Musculoskeletal and connective tissue disorders) | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 1 | 1
Skin Burning Sensation (Skin and subcutaneous tissue disorders) | 1 | 0
Skin Fissures (Skin and subcutaneous tissue disorders) | 0 | 1
Flushing (Vascular disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.